CLINICAL TRIAL: NCT01056224
Title: The Dose Effects of Remifentanil Boluses on the Hemodynamic Response to Skull Pin Insertion.
Brief Title: Effect of Remifentanil Boluses on Hemodynamics in Skull Pin Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Atul Prabhu, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-0684-B
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Skull Pin Insertion; Short Duration Analgesia
Keywords: skull pin insertion; remifentanil; short acting opioid; craniotomy; cervical spine surgery; hemodynamic changes; dose requirement; age related
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- 1.25 ug/kg normo-tensive 20-40 year olds (Experimental): A single bolus dose of 1.25 micrograms per kilogram body weight will be administered at the time of skull pin insertion in normo-tensive patients aged 20 to 40 years old.
  Interventions: Drug: Remifentanil
- 1.5 ug/kg normo-tensive 20-40 year olds (Experimental): A single bolus dose of 1.5 micrograms per kilogram body weight will be administered at the time of skull pin insertion in normo-tensive patients aged 20 to 40 years old.
  Interventions: Drug: Remifentanil
- 1.75 ug/kg normo-tensive 20-40 year olds (Experimental): A single bolus dose of 1.75 micrograms per kilogram body weight will be administered at the time of skull pin insertion in normo-tensive patients aged 20 to 40 years old.
  Interventions: Drug: Remifentanil
- 1 ug/kg normo-tensive 65-75 year olds (Experimental): A single bolus dose of 1 microgram per kilogram body weight will be administered at the time of skull pin insertion in normo-tensive patients aged 65 to 75 years old.
  Interventions: Drug: Remifentanil
- 1.25 ug/kg normo-tensive 65-75 year olds (Experimental): A single bolus dose of 1.25 micrograms per kilogram body weight will be administered at the time of skull pin insertion in normo-tensive patients aged 65 to 75 years old.
  Interventions: Drug: Remifentanil
- 1.5 ug/kg normo-tensive 65-75 year olds (Experimental): 1.5 ug/kg normo-tensive 65-75 year olds
  A single bolus dose of 1.5 micrograms per kilogram body weight will be administered at the time of skull pin insertion in normo-tensive patients aged 65 to 75 years old.
  Interventions: Drug: Remifentanil
- 1 ug/kg hyper-tensive 65-75 year olds (Experimental): A single bolus dose of 1 microgram per kilogram body weight will be administered at the time of skull pin insertion in hyper-tensive patients aged 65 to 75 years old.
  Interventions: Drug: Remifentanil
- 1.25 ug/kg hyper-tensive 65-75 year olds (Experimental): A single bolus dose of 1.25 micrograms per kilogram body weight will be administered at the time of skull pin insertion in hyper-tensive patients aged 65 to 75 years old.
  Interventions: Drug: Remifentanil
- 1.5 ug/kg hyper-tensive 65-75 year olds (Experimental): A single bolus dose of 1.5 micrograms per kilogram body weight will be administered at the time of skull pin insertion in hyper-tensive patients aged 65 to 75 years old.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — A single bolus dose of Remifentanil will be administered at the time of skull pin insertion

SUMMARY:
Skull pin insertion during craniotomies is a brief, intensely stimulating, painful stimuli occurring during the conduct of a neurosurgical or spine anesthetic. Remifentanil is an ultra short acting opioid that has been successfully used to blunt hemodynamic responses in a wide variety of clinical scenarios. It is our intention to ascertain the optimal dose for blunting the hemodynamic response to skull pin insertion using remifentanil.

DETAILED DESCRIPTION:
Skull pin insertion is commonly required for craniotomies and cervical spine surgery. It is a brief but highly stimulating maneuver performed following induction, during a period of light anesthesia, and may cause significant rise in blood pressure, heart rate and intracranial pressure if not anticipated and treated.

A wide variety of methods have been shown to be effective at blunting this hypertensive response. These include intravenous agents such as fentanyl, sufentanil, clonidine, ketamine and magnesium sulphate, local anesthetic methods such as injection at pin sites or full scalp blocks, deepening the volatile agent, oral premedication or a combination of these methods. There is no consensus on which of these methods is the best. Many anesthesiologists simply use boluses of propofol - a reliable way of accomplishing this effect with a familiar drug. It is also very common for anesthesiologists to use remifentanil, by increasing the infusion rate and or bolusing.

Remifentanil is an ultra-short acting opiate with such rapid onset and offset, that it is most easily and safely delivered by infusion. Increasingly in the literature, however, are reports of remifentanil administered as boluses rather than infusions. Boluses may be ideal for very short stimulating procedures such as intubation and skull pin fixation where a quick onset and offset are desired. Although the safety of bolusing remifentanil has been established in many studies , some authors are still apprehensive . Care must be taken to avoid bolusing with greater doses than required since this may lead to bradycardia and hypotension. In non-ventilated patients, respiratory depression is common and chest wall rigidity may occur at doses larger than 4ug/kg9.

Different bolus dose-effect studies have recommended the following for remifentanil in a variety of clinical settings:

* 3-5ug/kg with propofol 2mg/kg for intubation without muscle relaxants ,
* 2ug/kg with propofol TCI (>4ug/ml) and cisatracurium for intubation (no additional hemodynamic benefit using 4ug/kg)
* 1-1.25ug/kg for rapid sequence intubation with thiopentone 5-7mg/kg and succinylcholine 1mg/kg
* ED50 of 1.7ug/kg and ED95 of 2.88ug/kg for good to excellent intubating conditions in both infants and children (when used with 10ug/kg glycopyrrolate and 4mg/kg propofol)
* 3ug/kg (plus 4mg/kg propofol) provides similar intubating conditions when used in place of succinylcholine 2mg/kg for intubation in infants8

Remifentanil is not currently recommended for the following settings:

* As a sole agent for loss of consciousness with a high ED50 of 12ug/kg, lack of reliability and muscle rigidity common at such high doses
* Wide interindividual variability limit its use for labor analgesia (0.2-0.8ug/kg, median dose of 0.4ug/kg)

In neurosurgery, it is common to administer remifentanil as an infusion. Optimal infusion rates have already been investigated for intracranial surgery . However it is increasingly common to administer remifentanil as a bolus particularly during skull pin fixation, due to the desirable quick onset and offset, and there are no studies at present that have investigated optimal dose requirements for boluses in this setting.

At our institution we commonly administer remifentanil as a bolus during skull pin fixation and are interested in determining which bolus doses are safe and effective

ELIGIBILITY:
Inclusion Criteria:

Patients requiring skull pin fixation and general anesthesia for:

* Elective cervical spine surgery
* Elective craniotomies/brain tumor resection
* Elective transsphenoidal pituitary hypophysectomies

Exclusion Criteria:

Patients with evidence of raised intracranial pressure:

* GSC < 15
* Radiological evidence of significant rise in ICP (e.g. midline shift)
* Vascular anomalies in the brain

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To validate the safety and effectiveness of using remifentanil as a bolus for skull pin fixation | 10 minutes

SECONDARY OUTCOMES:
To determine the optimal doses for remifentanil in order to blunt the hemodynamic changes associated with skull pin fixation | 10 minutes
to assess variability in dose requirements of remifentanil | 10 minutes
to compare the dose effects in younger (20-40yo) vs. older (65-75yo) age groups | 10 minutes
to compare the dose effects in older (65-75yo) age groups in hypertensive versus non-hypertensive patients | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Atul Prabhu, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada